CLINICAL TRIAL: NCT02987569
Title: Teen Connections for Support From Multidisciplinary Professionals & Peers
Brief Title: Teen and Young Adult Connections for Support From Multidisciplinary Professionals & Peers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00004067; R01NR015743-01A1 (NIH)
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Short Bowel Syndrome; Malabsorption; Malnutrition
Keywords: Home Parenteral Nutrition; HPN; Total Parenteral Nutrition; TPN; mConnect; SBS; short bowel disorder; telehealth; telemedicine
MeSH Terms: conditions — Short Bowel Syndrome; Malabsorption Syndromes; Malnutrition; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group One (Experimental): Intervention
  Interventions: Behavioral: mConnect plus mobile connections to multidisciplinary professionals & peers
- Group Two (Active Comparator): Control
  Interventions: Behavioral: iPad use plus one mobile connections to multidisciplinary professionals & peers

INTERVENTIONS:
Behavioral: mConnect plus mobile connections to multidisciplinary professionals & peers — mConnect is the integration of evidence-based HPN interventions delivered via professionally moderated iPad visual meetings with peers, and reinforced by HPN related skill-building games (apps) and iPad music guided short naps.
  Arms: Group One
Behavioral: iPad use plus one mobile connections to multidisciplinary professionals & peers — iPad with a data plan and one professionally moderated iPad visual meeting with peers.
  Arms: Group Two

SUMMARY:
12 month study testing mobile delivery of health information and connections to professionals and peers to improve health of teen/young adult HPN users.

DETAILED DESCRIPTION:
This research study will test the effect of in-home/mobile HPN support delivered to teen and young adult home parenteral nutrition (HPN) patients and family members over handheld personal computers. Effects on health status, QoL, and fatigue will be assessed over time between groups of study subjects from the ages of 13 through 30 randomized to one of two groups. Group One (intervention group) will receive mConnect, integrated evidence-based interventions (skill-building games, restorative naps & peer support) via mobile iPad and Internet delivery plus two real-time audiovisual encrypted connections with multidisciplinary professionals and peers. Group Two (control group) will receive healthy activity information via mobile iPad and Internet delivery plus one real-time audiovisual encrypted connection with professionals and peers.

ELIGIBILITY:
Inclusion Criteria:

* Total parenteral nutrition (TPN) patients/users and family members/caregivers (defined as those individuals involved in daily home HPN care) age 13 and older
* TPN users (also called HPN users) ages 13 through 30 must be receiving intravenous nutrition for a non-malignant short bowel disorder
* Read, write, speak English and provide informed consent
* Be able to participate in group clinic visits

Exclusion Criteria:

* Enteral nutrition dependency only
* Less than 13 years of age
* 13 through 17 years of age without parental consent
* Currently enrolled in an intervention study or HPN management program
* Severe cognitive impairment
* Disability disorders (e.g. blindness which cannot be accommodated for active participation in the group clinics

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2016-07; Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Health Survey SF-12v2 (predicts future health services use). | T0 (baseline data collection)
  Physical and mental health status from each person's perspective. 7-Item Likert
Quality of Life (Cantril Ladder) | T0 (baseline data collection)
  Ratings of quality of life over time that are sensitive to changes in health. 3-Item Likert
Beck Depression Inventory-II (BDI-II) | T0 (baseline data collection)
  Assesses assess the intensity of depression into alignment with DSM-IV criteria. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression. 21-Item
Use of Healthy Living Activities Prompts, health intentions that predict engagement in targeted activities. | T2 (month 1-2/mConnect intervention period)
  Intention scale for healthy activities use (iPad discussion sessions, website use including games; mConnect use) 10-Item Likert
Use of Healthy Living Activities Prompts, health intentions that predict engagement in targeted activities. | T3 (month 3-4/mConnect intervention period)
  Intention scale for healthy activities use (iPad discussion sessions, website use including games; mConnect use) 10-Item Likert
Beck Depression Inventory-II (BDI-II) | T3 (4 months: change from T0/baseline)
  Assesses assess the intensity of depression into alignment with DSM-IV criteria. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression. 21-Item
Health Survey SF-12v2 (predicts future health services use). | T3 (4 months: change from T0/baseline)
  Physical and mental health status from each person's perspective. 7-Item Likert
Quality of Life (Cantril Ladder) | T3 (4 months: change from T0/baseline)
  Ratings of quality of life over time that are sensitive to changes in health. 3-Item Likert
Health Survey SF-12v2 (predicts future health services use). | T4 (8 months: change from T3/4 months)
  Physical and mental health status from each person's perspective. 7-Item Likert
Quality of Life (Cantril Ladder) | T4 (8 months: change from T3/4 months)
  Ratings of quality of life over time that are sensitive to changes in health. 3-Item Likert
Beck Depression Inventory-II (BDI-II) | T4 (8 months: change from T3/4 months)
  Assesses assess the intensity of depression into alignment with DSM-IV criteria. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression. 21-Item
Health Survey SF-12v2 (predicts future health services use). | T5 (12 months: change from T4/8 months)
  Physical and mental health status from each person's perspective. 7-Item Likert
Quality of Life (Cantril Ladder) | T5 (12 months: change from T4/8 months)
  Ratings of quality of life over time that are sensitive to changes in health. 3-Item Likert
Beck Depression Inventory-II (BDI-II) | T5 (12 months: change from T4/8 months)
  Assesses assess the intensity of depression into alignment with DSM-IV criteria. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression. 21-Item

SECONDARY OUTCOMES:
Preparedness (measures skills needed for independent HPN home care). | T0 (baseline data collection)
  Ability to manage home-care; low score = needs home care assistance. 8-Item Likert
COOPS Social Support Scale | T0 (baseline data collection)
  Ratings on having others who help, listen & provide tangible assistance support. 13-Item Likert
Preparedness (measures skills needed for independent HPN home care). | T3 (4 months: change from T0/baseline)
  Ability to manage home-care; low score = needs home care assistance. 8-Item Likert
COOPS Social Support Scale | T3 (4 months: change from T0/baseline)
  Ratings on having others who help, listen & provide tangible assistance support. 13-Item Likert
Mobile Care Helpfulness & Willingness-to-Pay Fees for Distance Health. | T4 (8 months)
  Rating of Helpfulness and willingness to pay for mobile care delivery. 10-Item Likert
Preparedness (measures skills needed for independent HPN home care). | T4 (8 months: change from T3/4 months)
  Ability to manage home-care; low score = needs home care assistance. 8-Item Likert
COOPS Social Support Scale | T4 (8 months: change from T3/4 months)
  Ratings on having others who help, listen & provide tangible assistance support. 13-Item Likert
Preparedness (measures skills needed for independent HPN home care). | T5 (12 months: change from T4/8 months)
  Ability to manage home-care; low score = needs home care assistance. 8-Item Likert
COOPS Social Support Scale | T5 (12 months: change from T4/8 months)
  Ratings on having others who help, listen & provide tangible assistance support. 13-Item Likert

CONTACTS AND LOCATIONS:
Overall Officials: Carol E Smith, RN, PhD, FAAN, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
All data is de-identified and will be reported only in aggregate.

REFERENCES:
- [Background] Nelson EL, Yadrich DM, Thompson N, Wright S, Stone K, Adams N, Werkowitch M, Smith CE. Telemedicine Support Groups for Home Parenteral Nutrition Users. Nutr Clin Pract. 2017 Dec;32(6):789-798. doi: 10.1177/0884533617735527. Epub 2017 Oct 10. PMID 29016235